CLINICAL TRIAL: NCT04732741
Title: Diagnostic Accuracy of Salivary Gamma-synuclein in Oral Malignant and Premalignant Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma mohamed saad-eldin mahmoud, Resident at the faculty of Dentistry, Cairo University
Other Study IDs: SS2021
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Oral Cancer; Oral Lichen Planus; Oral Leukoplakia; Premalignant Lesion
MeSH Terms: conditions — Mouth Neoplasms; Lichen Planus, Oral; Leukoplakia, Oral

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Salivary sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oral Cancer: patients diagnosed clinically and histopathologically with oral cancer who have yet to receive any treatment.
  Interventions: Diagnostic Test: Salivary Gamma-synuclein; Diagnostic Test: Incisional biopsy; Diagnostic Test: Conventional visual and tactile examination
- Premalignant lesions: patients diagnosed clinically and histopathologically with oral potentially malignant lesions who have not yet to receive treatment or had a month wash-out period from any previous treatment.
  Interventions: Diagnostic Test: Salivary Gamma-synuclein; Diagnostic Test: Incisional biopsy; Diagnostic Test: Conventional visual and tactile examination
- Control Group: healthy individuals who will be examined clinically through conventional visual and tactile examination to ensure no oral lesions are present and through thorough medical history
  Interventions: Diagnostic Test: Salivary Gamma-synuclein; Diagnostic Test: Conventional visual and tactile examination

INTERVENTIONS:
Diagnostic Test: Salivary Gamma-synuclein — Gamma-synuclein salivary levels measured using ELISA assay
Diagnostic Test: Incisional biopsy — A) Biopsy (reference standard): biopsy for group 1 will be performed by specialists in the national cancer institute.
  B) Biopsy for oral potentially malignant lesions will be performed by the candidate from the most representative region.
  Groups: Oral Cancer; Premalignant lesions
Diagnostic Test: Conventional visual and tactile examination — Conventional visual and tactile examination using light and mirror

SUMMARY:
Synucleins are a family of small, highly conserved proteins found in vertebrates and are specially abundant in neurons particularly in presynaptic terminals (Surguchov et al., 2001). Gamma-synuclein is the third member of the synuclein family, and is predominantly found in the cytosol of tumor cells and functions both intra- and extra-cellularly. It is involved in the pathogenesis of different types of cancer and some neurodegenerative diseases (Liu et al., 2018). Smoking - a major risk factor for oral cancer and its progression - and nicotine-containing products were found to time-dependently up-regulate the Gamma-synuclein expression in cancer cells (Hsu et al., 2020a).

Gamma-synuclein is released from tumor cells and was found to be elevated in tumors such as urinary bladder cancer (Liu et al., 2016), colorectal cancer, gastric adenocarcinomas and esophageal cancer (Liu et al., 2012). It is present in blood, serum, cerebrospinal fluid and saliva. The detection of extracellular synucleins in body fluids can reveal the first steps of the disease thus it can be used as a potential tool for early cancer detection (Surguchov, 2016).

This study aims to identify the diagnostic accuracy of Gamma-synuclein in differentiating between oral malignant lesions and oral premalignant lesions.

ELIGIBILITY:
Inclusion Criteria:

Group 1: patients with malignant lesions will be diagnosed through clinical and histopathological examination of tissue biopsy.

Group 2: patients with oral potentially malignant lesions will be diagnosed clinically and histopathological examination of tissue biopsy.

Group 3: healthy individuals who will be examined clinically through conventional visual and tactile examination to ensure no oral lesions are present and through thorough medical history

Exclusion Criteria:

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: patients with malignant lesions will be diagnosed through clinical and histopathological examination of tissue biopsy.
  Group 2: patients with oral potentially malignant lesions will be diagnosed clinically and histopathological examination of tissue biopsy.
  Group 3: healthy individuals who will be examined clinically through conventional visual and tactile examination to ensure no oral lesions are present and through thorough medical history
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2021-03-10 (Estimated); Primary Completion 2021-12-10 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
Gamma-synuclein level sensitivity and specificity | At same time as biopsy
  Measured using ELISA reader

IPD SHARING:
Plan to Share IPD: Undecided